CLINICAL TRIAL: NCT02078635
Title: The Canada-wide Human Nutrition Trialists' Network
Brief Title: Magnetic Resonance Imaging-Portfolio Diet Study #7
Acronym: MRIPD#7
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was amalgamated with another study to include exercise as another intervention.
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); Laval University (Other); University of Manitoba (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 13-260; FRN 129920 (Other Grant/Funding Number: Canadian Institutes of Health Research, Operating Grant)
Record Dates: First submitted 2014-02-18; First posted 2014-03-05 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Hypercholesterolemia; Diabetes; Metabolic Syndrome; Obesity
Keywords: Arterial plaque; portfolio diet; dietary modification; dietary trials; Canadian Network; knowledge synthesis and translation; Magnetic resonance imaging
MeSH Terms: conditions — Cardiovascular Diseases; Hypercholesterolemia; Diabetes Mellitus; Metabolic Syndrome; Obesity | interventions — Diet; Nutrition Assessment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Portfolio Plus Diet (Experimental): Participants will be advised to follow a low glycemic index dietary portfolio. Specifically, the advice will be to limit saturated fat (to <7% of total calories and cholesterol to <200 mg/d) plus inclusion of viscous fibres, soy protein, plant sterols and nuts, 5% extra monounsaturated fat and selection of low glycemic index foods; emphasizing current recommendations for fruit and vegetable intakes (5-10 servings/d)
  Interventions: Behavioral: Portfolio Plus Diet
- DASH-like (high fibre) diet (Active Comparator): The DASH-like dietary advice will emphasize a diet of whole grains, low-fat dairy and current recommendations for fruit and vegetables (5-10 servings/day)
  Interventions: Behavioral: DASH-like (high fibre) dietary advice

INTERVENTIONS:
Behavioral: Portfolio Plus Diet — Foods on the Portfolio Plus plan will contribute 9 g/1000 kcal viscous fibre as β-glucan (oats, barley, oat bran bread and soups) and psyllium (cereal), 1 g plant sterol/1000 kcal diet (in sterol margarine), 22.5 g soy protein/1000 kcal (soy burgers, dogs, links, other soy meat analogues, soy milks, yogurts and cheese) and additional sources of plant proteins from pulses (eg. lentils, chickpeas, beans, etc); and 22.5 g almonds or equivalent of other nuts/1000 kcal and increase MUFA (as olive and canola oils, avocados, nuts, margarine and salad dressings). The glycemic index will be reduced from 83 to 70 GI units (bread scale)
  Other Names: Dietary Portfolio of cholesterol-lowering foods; Enhanced portfolio; Portfolio eating plan
  Arms: Portfolio Plus Diet
Behavioral: DASH-like (high fibre) dietary advice — Dietary advice will be given to encourage intake of whole grain foods (brown rice, whole wheat breads, muffins and breakfast cereals); to reduce red meat consumption, choose low fat dairy foods and a control margarine
  Other Names: high fibre diet
  Arms: DASH-like (high fibre) diet

SUMMARY:
Presently in Canada, 29% of deaths are due to cardiovascular disease (CVD), costing $20.9 billion annually. The investigators have, therefore, brought together an unique network of investigators at different stages in their careers with a range of disciplines (nutrition, cardiology, diabetes, imaging, physics, clinical trials, statistics, laboratory medicine, primary care, genetics, psychology, knowledge translation (KT), and epidemiology) and with international recognition , experience and connections, to undertake a multi-centre study which will test the ability of the dietary Portfolio PLUS approach over 3 years to reduce the progression of plaque build-up in the carotid artery as assessed by Magnetic Resonance Imaging (MRI) in individuals with hypercholesterolemia.

The dietary portfolio of cholesterol-lowering foods (viscous fibres, soy protein, plant sterol and nuts) which has been proven in many of their studies to be an effective cholesterol-lowering diet will be further enhanced by increased levels of monounsaturated fats (MUFA) and low glycemic index foods. Will this enhanced dietary strategy (dietary Portfolio PLUS ) reduce the progression of carotid atheromatous lesions, LDL-C and blood pressure while reducing the number of hyperlipidemic individuals requiring statins?

DETAILED DESCRIPTION:
As Western populations age and as body weight increases, the need for dietary strategies to reduce Coronary Heart Disease (CHD) risk continues. The investigators are now in a position to put together a dietary approach which will be a significant advance over current dietary advice for CHD risk reduction. The investigators believe this study using imaging and functional techniques is now needed to 1) demonstrate an improvement in estimated CHD risk based on anatomical changes rather than serum risk factors. 2) encourage popular uptake and clinical use of this combination dietary strategy and 3) stimulate a larger longer term trial with CHD events.

Participants for this study will be recruited in 4 academic centres across Canada (Quebec, Toronto, Winnipeg and Vancouver). They will be in the low or moderate risk category based on the current Canadian Cardiovascular Society's (CCS) Guidelines 2012 and would normally be considered for initial treatment with lifestyle only. All participants will first be screened by ultrasound for the presence of plaque in the carotid arteries and will then be randomized to one of the 2 treatment arms: Portfolio Plus diet (test) or modified DASH diet (control), both given as routine clinical advice with follow up visits at 3-month intervals for 6 months and then twice yearly for the remainder of the 3 year trial.

Prior to starting either diet, participants will undergo screening ultrasound examination of both right and left carotids to enable selection of those individuals whose intima-media thickness would be 5-30% below the cut point considered by the Mannheim Consensus as relevant arterial thickening to ensure a relatively low risk group, yet with some measurable arterial thickening. The main outcome will be MRI assessment of maximum vessel wall volume. This assessment will be repeated at year 3. It will be emphasized at the outset that both the dietary portfolio and the DASH-like diets have been associated with benefits in terms of cholesterol reduction to provide equal encouragement for those randomized to the test and control groups. Portfolio and DASH-like dietary advice will consist of half hour individual sessions with the dietitian at baseline, 3, and 6 months and then at 6-month intervals. Prior to starting each diet, instruction will be given on achieving the dietary goals.

At follow-up visits, the participants' completed 7-day diet records will be discussed and the original advice reinforced. Every effort will be made to obtain study blood samples and carotid imaging data from all subjects at the designated times regardless of adherence to the dietary aspects of the study protocol. All subjects will be included in the intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants will be:

1. Adult males that are within 30% of their target LDL-cholesterol for the low or moderate risk category according to the 2012 Canadian Cardiovascular Society Guidelines.
2. Postmenopausal women that are within 30% of their target LDL-cholesterol for the low or moderate risk category according to the 2012 Canadian Cardiovascular Society Guidelines.

Participants will have the following characteristics:

* BMI 25-40 kg/m2 with body weight that has remained constant (within ±2kg) over the last 3 months preceding the onset of the study.
* Measurable arterial thickening at screening (carotid intima-media thickness of >1.0mm)
* Plus at least 1 of the following 3 criteria:

  * are treated with statins
  * are statin intolerant
  * have refused statin treatment after consultation with the appropriate physician

Exclusion Criteria:

Individuals with the following conditions will be excluded:

* major cardiovascular event

  * stroke or
  * myocardial infarction
* Cardiac conditions that compromise normal function

  * mitral valve disease
  * heart failure
  * angina
* familial hypercholesterolemia
* secondary causes of hypercholesterolemia

  * hypothyroidism (unless treated and on a stable dose of L-thyroxine)
  * renal or liver disease
* diabetes
* serum triglycerides >4.5 mmol/L
* uncontrolled blood pressure
* major disability
* disorders requiring continuous medical attention and treatment

  * chronic heart failure
  * liver disease
  * renal failure
  * cancer (except non-melanoma skin cancer--basal cell, squamous cell)
* chronic infections (bacterial or viral)
* chronic inflammatory diseases ( lupus, ulcerative colitis)
* other autoimmune diseases (eg celiac disease or gluten sensitivity)
* major surgery <6 months prior to randomization
* conditions that make them unsuitable for MRI (e.g. have metal implants or are claustrophobic)
* alcohol consumption >2 drinks/ day

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-10-07 (Actual); Study Completion 2014-10-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the maximum vessel wall volume of the carotid arteries | At baseline and year 3
  Assessed by MRI

SECONDARY OUTCOMES:
Intra-plaque hemorrhage (IPH) | At baseline and year 3
  Assessed by MRI
Intra-plaque lipid (lipid-rich necrotic core) | baseline and year 3
  Assessed by MRI
blood pressure and pulse rate | At months 0, 3, 6, 12, 18, 24, 30, 36
initiation of statin therapy | baseline and year 3
  According to current CCS guidelines

OTHER OUTCOMES:
LDL-cholesterol | At months, 0, 3, 6, 12, 18, 24, 30, 36
HDL-cholesterol | months 0, 3, 6, 12, 18, 24, 30, 36
C-reactive protein (CRP) | At months 0, 12, 24, and 36
The Medical Outcomes Study 36-Item Short Form Questionnaire (SF-36) | Months 0 and 36
  Survey on quality of life.
Genetic whole genome testing | month 0
  One time sample collection of buffy coat white cells for future analysis
satiety of the test and control diet | Months 0, 3, 6, 12, 18, 24, 30, 36
  Participants will assess their level of satiety on the test/control diet at each visit using a 9-point bipolar semantic scale ranging from -4 (being starved/ feeling weak and faint with hunger) to +4 (being Painfully full) with 0 being neutral (ie don't mind eating a little more or less).
Palatability of the test / control diets | Months 3, 6, 12, 18, 24, 30, and 36
  The palatability of the diet will by measured using a numerical scale of 1 to 10 (1= strongly dislike and 10 = like very much).

CONTACTS AND LOCATIONS:
Overall Officials: David J Jenkins, MD, Principal Investigator — St. Michael's Hospital / University of Toronto; Benoit Lamarche, PhD, Study Director — Laval University; Peter Jones, PhD, Study Director — University of Manitoba; Jiri Frohlich, MD, Study Director — University of British Columbia
Locations (4):
- Canada (4):
  - Healthy Heart Lipid Clinic, St. Paul's Hospital, Vancouver, British Columbia
  - Richardson Center for Functional Foods and Nutraceuticals and the St. Boniface Hospital Cardiovascular Center, University of Manitoba, Winnipeg, Manitoba
  - Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario
  - Institute of Nutraceuticals and Functional Foods and the Quebec Heart and Lung Institute, Laval University, Québec, Quebec

REFERENCES:
- [Background] Jenkins DJ, Jones PJ, Lamarche B, Kendall CW, Faulkner D, Cermakova L, Gigleux I, Ramprasath V, de Souza R, Ireland C, Patel D, Srichaikul K, Abdulnour S, Bashyam B, Collier C, Hoshizaki S, Josse RG, Leiter LA, Connelly PW, Frohlich J. Effect of a dietary portfolio of cholesterol-lowering foods given at 2 levels of intensity of dietary advice on serum lipids in hyperlipidemia: a randomized controlled trial. JAMA. 2011 Aug 24;306(8):831-9. doi: 10.1001/jama.2011.1202. PMID 21862744
- [Background] Statistics Canada. Mortality, Summary list of Causes 2008. Released October 18, 2011
- [Background] Conference Board of Canada. The Canadian Heart Healthy Strategy: Risk Factors and Future Cost Implications. Report of February 2010.
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Krauss RM, Eckel RH, Howard B, Appel LJ, Daniels SR, Deckelbaum RJ, Erdman JW Jr, Kris-Etherton P, Goldberg IJ, Kotchen TA, Lichtenstein AH, Mitch WE, Mullis R, Robinson K, Wylie-Rosett J, St Jeor S, Suttie J, Tribble DL, Bazzarre TL. AHA Dietary Guidelines: revision 2000: A statement for healthcare professionals from the Nutrition Committee of the American Heart Association. Circulation. 2000 Oct 31;102(18):2284-99. doi: 10.1161/01.cir.102.18.2284. No abstract available. PMID 11056107
- [Background] Genest J, McPherson R, Frohlich J, Anderson T, Campbell N, Carpentier A, Couture P, Dufour R, Fodor G, Francis GA, Grover S, Gupta M, Hegele RA, Lau DC, Leiter L, Lewis GF, Lonn E, Mancini GB, Ng D, Pearson GJ, Sniderman A, Stone JA, Ur E. 2009 Canadian Cardiovascular Society/Canadian guidelines for the diagnosis and treatment of dyslipidemia and prevention of cardiovascular disease in the adult - 2009 recommendations. Can J Cardiol. 2009 Oct;25(10):567-79. doi: 10.1016/s0828-282x(09)70715-9. PMID 19812802
- [Background] Ornish D, Brown SE, Scherwitz LW, Billings JH, Armstrong WT, Ports TA, McLanahan SM, Kirkeeide RL, Brand RJ, Gould KL. Can lifestyle changes reverse coronary heart disease? The Lifestyle Heart Trial. Lancet. 1990 Jul 21;336(8708):129-33. doi: 10.1016/0140-6736(90)91656-u. PMID 1973470
- [Background] Atkins R. Dr. Atkins' New Diet Revolution. New York NAB.
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Jenkins DJ, Chiavaroli L, Wong JM, Kendall C, Lewis GF, Vidgen E, Connelly PW, Leiter LA, Josse RG, Lamarche B. Adding monounsaturated fatty acids to a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. CMAJ. 2010 Dec 14;182(18):1961-7. doi: 10.1503/cmaj.092128. Epub 2010 Nov 1. PMID 21041432
- [Background] Food labeling: health claims; plant sterol/stanol esters and coronary heart disease. Food and Drug Administration, HHS. Interim final rule. Fed Regist. 2000 Sep 8;65(175):54686-739. PMID 11503640
- [Background] Jenkins DJ, Kendall CW, McKeown-Eyssen G, Josse RG, Silverberg J, Booth GL, Vidgen E, Josse AR, Nguyen TH, Corrigan S, Banach MS, Ares S, Mitchell S, Emam A, Augustin LS, Parker TL, Leiter LA. Effect of a low-glycemic index or a high-cereal fiber diet on type 2 diabetes: a randomized trial. JAMA. 2008 Dec 17;300(23):2742-53. doi: 10.1001/jama.2008.808. PMID 19088352
- [Background] Jenkins DJ, Kendall CW, Augustin LS, Mitchell S, Sahye-Pudaruth S, Blanco Mejia S, Chiavaroli L, Mirrahimi A, Ireland C, Bashyam B, Vidgen E, de Souza RJ, Sievenpiper JL, Coveney J, Leiter LA, Josse RG. Effect of legumes as part of a low glycemic index diet on glycemic control and cardiovascular risk factors in type 2 diabetes mellitus: a randomized controlled trial. Arch Intern Med. 2012 Nov 26;172(21):1653-60. doi: 10.1001/2013.jamainternmed.70. PMID 23089999
- [Background] Jones PJ, AbuMweis SS. Phytosterols as functional food ingredients: linkages to cardiovascular disease and cancer. Curr Opin Clin Nutr Metab Care. 2009 Mar;12(2):147-51. doi: 10.1097/mco.0b013e328326770f. PMID 19209468
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Background] Jenkins DJ, Kendall CW, Faulkner D, Vidgen E, Trautwein EA, Parker TL, Marchie A, Koumbridis G, Lapsley KG, Josse RG, Leiter LA, Connelly PW. A dietary portfolio approach to cholesterol reduction: combined effects of plant sterols, vegetable proteins, and viscous fibers in hypercholesterolemia. Metabolism. 2002 Dec;51(12):1596-604. doi: 10.1053/meta.2002.35578. PMID 12489074
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner D, Vidgen E, Lapsley KG, Trautwein EA, Parker TL, Josse RG, Leiter LA, Connelly PW. The effect of combining plant sterols, soy protein, viscous fibers, and almonds in treating hypercholesterolemia. Metabolism. 2003 Nov;52(11):1478-83. doi: 10.1016/s0026-0495(03)00260-9. PMID 14624410
- [Background] Jenkins DJ, Wolever TM, Taylor RH, Barker H, Fielden H, Baldwin JM, Bowling AC, Newman HC, Jenkins AL, Goff DV. Glycemic index of foods: a physiological basis for carbohydrate exchange. Am J Clin Nutr. 1981 Mar;34(3):362-6. doi: 10.1093/ajcn/34.3.362. PMID 6259925
- [Background] Hu FB, Stampfer MJ, Manson JE, Rimm EB, Colditz GA, Rosner BA, Speizer FE, Hennekens CH, Willett WC. Frequent nut consumption and risk of coronary heart disease in women: prospective cohort study. BMJ. 1998 Nov 14;317(7169):1341-5. doi: 10.1136/bmj.317.7169.1341. PMID 9812929
- [Background] Liu S, Willett WC, Stampfer MJ, Hu FB, Franz M, Sampson L, Hennekens CH, Manson JE. A prospective study of dietary glycemic load, carbohydrate intake, and risk of coronary heart disease in US women. Am J Clin Nutr. 2000 Jun;71(6):1455-61. doi: 10.1093/ajcn/71.6.1455. PMID 10837285
- [Background] Pereira MA, O'Reilly E, Augustsson K, Fraser GE, Goldbourt U, Heitmann BL, Hallmans G, Knekt P, Liu S, Pietinen P, Spiegelman D, Stevens J, Virtamo J, Willett WC, Ascherio A. Dietary fiber and risk of coronary heart disease: a pooled analysis of cohort studies. Arch Intern Med. 2004 Feb 23;164(4):370-6. doi: 10.1001/archinte.164.4.370. PMID 14980987
- [Background] Mensink RP, Zock PL, Kester AD, Katan MB. Effects of dietary fatty acids and carbohydrates on the ratio of serum total to HDL cholesterol and on serum lipids and apolipoproteins: a meta-analysis of 60 controlled trials. Am J Clin Nutr. 2003 May;77(5):1146-55. doi: 10.1093/ajcn/77.5.1146. PMID 12716665
- [Background] Keys A, Aravanis C, Blackburn HW, Van Buchem FS, Buzina R, Djordjevic BD, Dontas AS, Fidanza F, Karvonen MJ, Kimura N, Lekos D, Monti M, Puddu V, Taylor HL. Epidemiological studies related to coronary heart disease: characteristics of men aged 40-59 in seven countries. Acta Med Scand Suppl. 1966;460:1-392. No abstract available. PMID 5226858
- [Background] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428
- [Background] Touboul PJ, Hennerici MG, Meairs S, Adams H, Amarenco P, Desvarieux M, Ebrahim S, Fatar M, Hernandez Hernandez R, Kownator S, Prati P, Rundek T, Taylor A, Bornstein N, Csiba L, Vicaut E, Woo KS, Zannad F; Advisory Board of the 3rd Watching the Risk Symposium 2004, 13th European Stroke Conference. Mannheim intima-media thickness consensus. Cerebrovasc Dis. 2004;18(4):346-9. doi: 10.1159/000081812. Epub 2004 Nov 2. PMID 15523176
- [Background] Jenkins DJ, Kendall CW, Faulkner DA, Nguyen T, Kemp T, Marchie A, Wong JM, de Souza R, Emam A, Vidgen E, Trautwein EA, Lapsley KG, Holmes C, Josse RG, Leiter LA, Connelly PW, Singer W. Assessment of the longer-term effects of a dietary portfolio of cholesterol-lowering foods in hypercholesterolemia. Am J Clin Nutr. 2006 Mar;83(3):582-91. doi: 10.1093/ajcn.83.3.582. PMID 16522904
- [Background] The DASH diet. Dietary Approaches to Stop Hypertension. Lippincotts Prim Care Pract. 1998 Sep-Oct;2(5):536-8. No abstract available. PMID 9791393
- [Background] Murie-Fernandez M, Irimia P, Toledo E, Martinez-Vila E, Buil-Cosiales P, Serrano-Martinez M, Ruiz-Gutierrez V, Ros E, Estruch R, Martinez-Gonzalez MA; PREDIMED Investigators. Carotid intima-media thickness changes with Mediterranean diet: a randomized trial (PREDIMED-Navarra). Atherosclerosis. 2011 Nov;219(1):158-62. doi: 10.1016/j.atherosclerosis.2011.06.050. Epub 2011 Jul 6. PMID 21802081
- [Background] Black AE, Goldberg GR, Jebb SA, Livingstone MB, Cole TJ, Prentice AM. Critical evaluation of energy intake data using fundamental principles of energy physiology: 2. Evaluating the results of published surveys. Eur J Clin Nutr. 1991 Dec;45(12):583-99. PMID 1810720
- [Background] Bingham SA, Gill C, Welch A, Day K, Cassidy A, Khaw KT, Sneyd MJ, Key TJ, Roe L, Day NE. Comparison of dietary assessment methods in nutritional epidemiology: weighed records v. 24 h recalls, food-frequency questionnaires and estimated-diet records. Br J Nutr. 1994 Oct;72(4):619-43. doi: 10.1079/bjn19940064. PMID 7986792
- [Background] Composition of Foods, Agriculture Handbook No. 8. In: Agriculture UDo, ed.: The Agriculture Research Service, 1992.
- [Background] Smilde TJ, van Wissen S, Wollersheim H, Kastelein JJ, Stalenhoef AF. Genetic and metabolic factors predicting risk of cardiovascular disease in familial hypercholesterolemia. Neth J Med. 2001 Oct;59(4):184-95. doi: 10.1016/s0300-2977(01)00155-3. PMID 11578794
- [Background] van Wissen S, Smilde TJ, Trip MD, Stalenhoef AF, Kastelein JJ. Long-term safety and efficacy of high-dose atorvastatin treatment in patients with familial hypercholesterolemia. Am J Cardiol. 2005 Jan 15;95(2):264-6. doi: 10.1016/j.amjcard.2004.09.015. PMID 15642565
- [Background] Johnsen SH, Mathiesen EB, Joakimsen O, Stensland E, Wilsgaard T, Lochen ML, Njolstad I, Arnesen E. Carotid atherosclerosis is a stronger predictor of myocardial infarction in women than in men: a 6-year follow-up study of 6226 persons: the Tromso Study. Stroke. 2007 Nov;38(11):2873-80. doi: 10.1161/STROKEAHA.107.487264. Epub 2007 Sep 27. PMID 17901390
- [Background] Mathiesen EB, Johnsen SH, Wilsgaard T, Bonaa KH, Lochen ML, Njolstad I. Carotid plaque area and intima-media thickness in prediction of first-ever ischemic stroke: a 10-year follow-up of 6584 men and women: the Tromso Study. Stroke. 2011 Apr;42(4):972-8. doi: 10.1161/STROKEAHA.110.589754. Epub 2011 Feb 10. PMID 21311059
- [Background] Spence JD. Technology Insight: ultrasound measurement of carotid plaque--patient management, genetic research, and therapy evaluation. Nat Clin Pract Neurol. 2006 Nov;2(11):611-9. doi: 10.1038/ncpneuro0324. PMID 17057748
- [Background] Saam T, Kerwin WS, Chu B, Cai J, Kampschulte A, Hatsukami TS, Zhao XQ, Polissar NL, Neradilek B, Yarnykh VL, Flemming K, Huston J 3rd, Insull W Jr, Morrisett JD, Rand SD, DeMarco KJ, Yuan C. Sample size calculation for clinical trials using magnetic resonance imaging for the quantitative assessment of carotid atherosclerosis. J Cardiovasc Magn Reson. 2005;7(5):799-808. doi: 10.1080/10976640500287703. PMID 16353440
- [Background] Lee GA. Determinants of quality of life five years after coronary artery bypass graft surgery. Heart Lung. 2009 Mar-Apr;38(2):91-9. doi: 10.1016/j.hrtlng.2008.04.003. Epub 2008 Sep 19. PMID 19254627
- [Background] Pischke CR, Weidner G, Elliott-Eller M, Ornish D. Lifestyle changes and clinical profile in coronary heart disease patients with an ejection fraction of <or=40% or >40% in the Multicenter Lifestyle Demonstration Project. Eur J Heart Fail. 2007 Sep;9(9):928-34. doi: 10.1016/j.ejheart.2007.05.009. Epub 2007 Jun 14. PMID 17572148